CLINICAL TRIAL: NCT02615652
Title: The Impact of Lifestyle on Mental Health Among Young Men in the Gilgel Gibe Field Research Center, Ethiopia: Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Konstanz (Other)
Collaborators: Jimma University (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Michael Odenwald, Researcher, Akademischer Rat, University of Konstanz
Other Study IDs: University of Konstanz
Record Dates: First submitted 2015-11-22; First posted 2015-11-26 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Common Mental Disorders (CMD); Psychotic Symptoms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Immunoassay test for the screening of khat alkaloids in urine.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: no intervention — no intervention, observational study

SUMMARY:
Researchers of the three collaborating universities implement a pilot observational study in "Gilgel Gibe Field Research Center", a health and demographic surveillance system run by the Jimma University, Ethiopia. In this setting, the investigators plan to study risk factors in young men for the development of common mental disorders and psychotic symptoms and the stability of distinct symptoms of mental disorders in the community. The investigators will explore in particular the impact of lifestyle on mental health in young men, including the traditional habit of chewing khat leaves, which contain amphetamine-like cathinone. Furthermore, the investigators want to demonstrate the reliability and validity of assessments performed by trained local interviewers.

ELIGIBILITY:
Inclusion Criteria:

* Male, Age 18 - 30, permanent residents in Gilgel Gibe

Exclusion Criteria:

* Prior existing severe mental health problems

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adult male inhabitants of the Gilgel Gibe field research center.
Sampling Method: Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
psychotic symptoms | through study completion, within 2 months
  presence of self-reported psychotic symptoms during the month before interview
symptoms of Common Mental Disorders | through study completion, within 2 months
  presence of self-reported CMD symptoms during the month before interview

SECONDARY OUTCOMES:
amount of khat use | through study completion, within 2 months
  self-reported amount of khat standard units consumed last week
amount of alcohol use | through study completion, within 2 months
  self-reported amount of alcohol standard units consumed last week